CLINICAL TRIAL: NCT04219605
Title: Evaluation of a Rapid Microscopic Diagnostic System for Different Vaginitis Conditions
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0120-19-COM1
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Bacterial Vaginosis; Candida Albicans Vulvovaginitis; Candida Vulvovaginitis; Trichomonas Vaginitis; Atrophic Vaginitis; Desquamative Inflammatory Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Trichomonas Vaginitis; Atrophic Vaginitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptomatic vaginitis patients: Symptomatic patients evaluated in the clinic for vulvovaginal symptoms.

SUMMARY:
Evaluate the diagnostic performance of the Gyni™ device to detect different vaginitis conditions by comparison to microscopic diagnosis and related lab tests.

DETAILED DESCRIPTION:
During gynecological exams, vaginal discharge samples will be are taken for testing the pH level, microscopic examination and laboratory examinations (vaginal cultures and sexually transmitted infections).

One additional sample will be taken intended for the Gyni™ system diagnosis. This additional examination will be performed in the clinic by pulling the cytobrush through a dedicated cartridge and scanning it in the Gyni table-top scanner. The result diagnosis will be anonymously kept in the cloud.

The diagnosis suggested by the Gyni system will not be visible to the physician in order to prevent any bias. Results from the physician, from the device and from the lab will be summarized and compared by the chief investigator

ELIGIBILITY:
Inclusion Criteria:

* Women with vaginal complaints: Discharge, Malodor, Itching, Irritation, Dyspareunia, Pain
* Age >= 18y

Exclusion Criteria:

* Age < 18y
* Not eligible to sign an informed consent
* Vaginal discharge samples found microscopically not interpret-able by the investigator due to patient using vaginal creams, ointments, lubricants or sperm presence.
* During menstruation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study examine a diagnostic test for vaginal inflammations (vaginitis) which is only applicable to female patients.
Study Population: Patients with vulvovaginal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance | 12 months
  Specificity and sensitivity of the device performance in regard to vaginitis conditions

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ben Chetrit, MD, Principal Investigator — Clalit HMO
Locations (1):
- Clalit HMO, Jerusalem, Jerusalem, Israel

REFERENCES:
- [Background] Lev-Sagie A, Strauss D, Ben Chetrit A. Diagnostic performance of an automated microscopy and pH test for diagnosis of vaginitis. NPJ Digit Med. 2023 Apr 13;6(1):66. doi: 10.1038/s41746-023-00815-w. PMID 37055473